CLINICAL TRIAL: NCT01802294
Title: Sinovuyo Caring Families Project - Pilot Randomised Controlled Trial of a Parenting Program to Reduce Child Behavior Problems in Xhosa Children Ages 3 to 8 in South Africa
Brief Title: Sinovuyo Caring Families Project - Pilot Trial
Acronym: SCFP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: University of Oxford (Other); Bangor University (Other); Ilifa Labantwana (Unknown)
Responsible Party: Principal Investigator, Dr Catherine L. Ward, Principal Investigator, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Griffin39
Record Dates: First submitted 2013-02-15; First posted 2013-03-01 (Estimated); Last update posted 2014-06-13 (Estimated); Status verified 2014-06

CONDITIONS: Child Behavior; Parenting; Child Abuse
Keywords: Randomized Controlled Trials as Topic; Child; Parents
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Parenting Program (Experimental): 12-week group-based parenting program (Sinovuyo Caring Family Programme) delivered in weekly sessions. Program is manualized.
  Interventions: Behavioral: Parenting Program
- Wait-list control (No Intervention): Wait-list control group. Program delivered 3 months after posttest.

INTERVENTIONS:
Behavioral: Parenting Program — Goal of the program is reduction in child behavior problems in high-risk South African families. Program will be delivered to caregivers responsible for the wellbeing of the child.
  Program activities will be delivered over 12 weekly group sessions with additional individualized in-home sessions. The groups (n = 15 participants per group) will meet weekly with community facilitators (n = 2 per group). Parenting skills will be developed during the sessions through role-plays, group-discussion, storytelling, and home practice activities.
  The program is manualized in isiXhosa.
  Other Names: Sinovuyo Caring Families Programme
  Arms: Parenting Program

SUMMARY:
This pilot feasibility trial will evaluate the Sinovuyo Caring Families Program in a small-scale randomized controlled trial in Cape Town, South Africa (n=60 families). The pilot study will use a mixed-methods approach to intervention evaluation. Self-report and observed quantitative data for intervention and control groups will be collected at pre-test and post-test evaluation. Primary outcomes will include parent-reports and observations of child behavior problems. In addition, as an exploratory study, this phase will examine initial pre-post intervention effects for potential mediating factors of parenting behavior, parental stress, parental depression, and perceived social support. However, this phase will not test mediation effects due to small sample sizes. Quantitative assessments will also collect data on program fidelity, exposure/adherence, participant engagement, and satisfaction. Furthermore, qualitative focus groups with intervention participants and group leaders will examine issues of program feasibility, content, deliver, and satisfaction. Randomization will be done on an individual level and include a wait-list control group that will receive the intervention 3 months after the post-test evaluation. Results from the feasibility pilot study will be shared with intervention partners and advisory groups. If necessary, final program adjustments will be made prior to further testing. Results will also be disseminated to community forums, local organizations, government stakeholders, and via academic conferences.

Research hypotheses:

Hypothesis 1: Children in the intervention group will demonstrate reduced observed and parent-reported child behavior problems in comparison to the control group.

Hypothesis 2: Parents in the intervention group will demonstrate increased observed and self-reported positive parenting outcomes and decreased observed and self-reported harsh and inconsistent parenting outcomes in comparison to the control group.

Hypothesis 3: Parents in the intervention group will demonstrate decreased parental depression and parental stress outcomes and increased perceived social support outcomes in comparison to the control group.

Hypothesis 4: The Sinovuyo Caring Families Program will be implemented with an acceptable degree of program fidelity, exposure/adherence, and participant satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* isiXhosa-speaking adults above the age of 18
* primary guardians of children aged 3-8 from Khayelitsha, Cape Town
* reside in the same household as child for at least 4 nights per week
* Score 11 or more on Eyberg Child Behavior Inventory Problem Scale

Exclusion Criteria:

* Severe mental health problems on Beck Depression Inventory
* Evidence of severe child maltreatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2013-02; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Eyberg Child Behavior Inventory | Change from baseline to 1 week post-program (13 weeks from baseline)
  This 36-item examines externalizing behavior problems in children ages 2 to 16 using both an Intensity Scale and Problem Scale. Parents are asked how often a specific behavior occurs and whether the behavior is considered a problem. Based on the most typical child behavior problems, items include "has poor table manners," "acts defiant when told to do something," "physically fights with sisters and brothers," and "fails to finish tasks or project." The Intensity Scale rates frequency of occurrence based on a 7-point Likert scale (1 = never occurs to 7 = always occurs). The Problem Scale measures whether the parent identifies a specific behavior as a problem (0 = no; 1 = yes). Both scales are summed up to create a total Intensity Score and Problem Score. Clinical cut-off scores suggested for psychopathological problem behavior are 131 for the Intensity Score and 11 for the Problem Score (Eyberg, 1999).
Family Observation Scale, 6th Edition | Change from baseline to 1 week post-program (13 weeks from baseline)
  The FOS-6 measures both consistency and intensity of child and parent behavior. Coding systems use a Likert scale from 0-4 to record whether and how often a particular behavior occurred (0 = behavior did not occur and/or was of low intensity; 4 = occurred a lot and/or was of high intensity). Codes are identified according to different behavioral categories through global and interval coding. Observed parent behavior includes harsh parenting, lax parenting, and praise. Similarly, child behaviors are non-compliance, proactive oppositionality, complaint, and withdrawal. Frequency and intensity scores are calculating by summing the individual scores and then dividing by the total number of observation intervals. Final scores are then calculated from means to generate an overall rating as well as for each subscale (Sanders, 2000).

SECONDARY OUTCOMES:
Parent-Child Conflict Tactics Scale (CTSPC) (Straus et al., 1998) | Change from baseline to 1 week post-program (13 weeks from baseline)
  The CTSPC (27-items) contains subscales measuring psychological aggression (5-items, e.g. - "shouted, yelled, or screamed at"), physical assault (13-items, e.g. - "hit on the bottom with a belt"), and neglect (5-items, e.g. - "were too drunk to take care of your child") as well as nonviolent discipline (4-items, e.g. - "explained why something was wrong"). Parents respond according to a Likert scale based on the number of times in the past 3 months each activity occurs (1 = never to 5 = three or more times). The CTSPC produces an overall harsh parenting score as well as for each subscale by summing the responses. It also measures the prevalence of harsh parenting by creating a dichotomized variable (0 = never, 1 = all other responses).
Parenting Young Children Scale (PARYC) | Change from baseline to 1 week post-program (13 weeks from baseline)
  The PARYC (14-items) measures the occurrence of specific parental behavior towards children (e.g. - "notice and praise your child's good behavior") during the previous month on a 7-point Likert scale (0 = never, 7 = almost daily), as well as whether performing this behaviour is currently a problem or difficult (0 = no, 1 = yes). Items are summed to create total frequency and problem scores, as well as for each subscale.
Parenting Stress Index-Short Form, Distress Subscale | Change from baseline to 1 week post-program (13 weeks from baseline)
  The Parenting Distress subscale (12-items) rates parents' responses on a 5-point Likert scale regarding the frequency of stress related to parenting within the past 3 months (1 = Never; 5 = Always). Items include parenting stress due to marital conflict (e.g. - "taking care of children causes problems between me and my spouse"), sense of parental competence (e.g. - "I feel inadequate as a parent"), and lack of support (e.g. - "I feel alone and without friends"). Items are summed to create a total score.
Beck Depression Inventory (BDI-II) | Change from baseline to 1 week post-program (13 weeks from baseline)
  The BDI-II is a 21-item scale designed to assess the intensity of depression in both clinical patients and for the general population. Respondents are asked to choose from a series of statements describing various symptoms on a four-point scale (e.g. - "Sadness: 0 = I do not feel sad; 1 = I feel sad much of the time; 2 = I am sad all the time; 3 = I am so sad or unhappy that I can't stand it"). Responses are then summed ranging from 0 to 63, with higher scores indicating higher levels of depressive symptoms. Recommended cut-off scores are 0-13 for minimal depression, 14-19 for mild depression, 20-28 for moderate depression, and 29-63 for severe depression (Beck, 1996).
Multidimensional Scale of Perceived Social Support (MSPSS, 12-items) | Change from baseline to 1 week post-program (13 weeks from baseline)
  Participants report on the levels of perceived social support based on a Likert scale of 1 to 7 (1 = very strongly disagree; 1 = very strongly agree). The MSPSS includes subscales for family support (e.g. - "I get the emotional support and help I need from my family"), friend support (e.g. - "I can count on my friends when things go wrong"), and other support (e.g. - "there is a special person who is around when I am in need"). Responses are summed to create subscale and total scores from 12 to 84 with higher scores indicating higher levels of perceived social support.
Parental Monitoring | Change from baseline to 1 week post-program (13 weeks from baseline)
  6-item subscale measuring parental monitoring from the Parenting Children and Adolescents Scale
Empathy and Personality traits of child | Baseline
  Two parent-report measures will be used to assess empathy and personality traits associated with a lack of empathy in children. Using Beatty and Willis (2007) 'probing based' paradigm, cognitive interviews will be conducted with some of the parents to assess understanding and the basis of responses, while a Theory of Mind battery will be administered to assess a child's theory of mind.
Theory of mind | Baseline
  The UCT Theory of Mind (ToM) battery developed by Hoogenhout and Malcolm-Smith (2014) is an adaption of the battery used by Steele and colleagues (2003). The measure consists of 11 ToM tasks that are divided into four modules of increasing difficulty (Early, Basic, Intermediate, and Advanced). The Early module assesses the ability to engage in pretend play and to understand other's desires, while the Basic module includes the assessment of the classic first-order false belief task (Baron-Cohen, Leslie & Frith, 1985; Wimmer & Perner, 1983). The Intermediate and Advanced modules include second-order false belief and the child's ability to recognize faux pas, sarcasm, irony, and to distinguish between lies and jokes respectively.
Cognitive status | Baseline
  The Grover-Counter Scale of Cognitive Development, designed to assess cognitive functioning, was initially developed for use with handicapped subjects and specifically where verbal communication between tester and testee is compromised. This makes the test appropriate for use where tester and testee's first language differ. The scale is based on Piagetian theory and associates each stage of the test with Piaget's stages of development. Minimum achievement cut-offs are specified for each stage. Provisional norms were established based on a convenience sample of normal African-language speaking children (3-10yrs).

OTHER OUTCOMES:
Implementation Fidelity | Measured weekly over the 12 weeks of the program
  In this pilot study, implementation fidelity will be measured using group leader self-report checklists to examine the extent to which core intervention components are delivered. These checklists will include specific activities for each session, such as home practice discussion and role-playing exercises. They will also measure the extent to which core parenting program theoretical concepts - such as child-led play, specific praise and encouragement, and the use of time-out - are implemented. Additionally, the research team will perform periodic observational assessments (4 per group) to verify the group leaders' self-report checklists.
Program exposure, adherence, and engagement | Measured weekly over the 12 weeks of the program
  Participation attendance registers for each session will assess exposure of participants to the intervention components. Furthermore, weekly self-report activity checklists based on a Likert scale of 1-4 (1 = none of the time, 4 = all of the time) will measure the extent to which participants actively engage with program components such as home practice activities (Glasgow et al., 1999). Finally, at the end of the program, qualitative focus groups will explore participants' experiences and the barriers to program exposure, adherence, and engagement.
Participant Satisfaction | Measured weekly over the 12 weeks of the program
  Participants will complete weekly evaluations (7-items) examining satisfaction of session content, activities, facilitator teaching, and group discussion. Participant satisfaction surveys of the overall program (40-items total) will investigate parents' perceptions of whether the program fulfilled their expectations (10-items), acceptability of delivery and teaching methods (10-items), acceptability of theoretical parenting techniques (10-items), and evaluation of program facilitators (5-items per facilitator). Reponses for weekly and overall surveys will be based on a Likert scale of 1 to 5 (e.g. - 1 = very unhelpful, 5 = very helpful). Items will be summed to create weekly satisfaction scores and an overall program satisfaction score.
Program feasibility | Measured immediately after the program is over (13 weeks from baseline)
  The feasibility pilot study will conduct qualitative focus groups with intervention participants (n = 15 participants per group, 2 groups) and in-depth interviews with the community health workers and program mentors (n = 4 facilitators, n = 2 mentors) in order to explore program acceptability. These will occur during the post-evaluation and examine the following themes: 1) participants' observed change in parenting practices and child behavior at home during the program; 2) acceptability and appropriateness of program materials, delivery, and key program components; and 3) existing barriers to participation during sessions and engagement in home practice and other activities. Interviews will also explore facilitators' challenges in implementing the program.
Revised Conflict Tactics Short Form | Change from baseline to 1 week post-program (13 weeks from baseline)
  The Revised Conflict Tactics Short Form scale (CTS2S; 10 items) measures exposure to intimate partner physical and psychological violence (Straus, 2004). Adapted from the Revised Conflict Tactics (CTS2) scale (Straus et al., 1996), the measurement uses adult self-report on the frequency of negotiation, physical assault, psychological aggression, sexual coercion, and physical injury. Answers are coded on a Likert scale of 0 to 3 (0 = never happened; 3 = more than 3 times in the past year) with an additional response of 7 for incidences that happened more than a year ago. The CTS2S measures overall indication of intimate partner violence on a level of severity (sum of items) and p
World Health Organization Alcohol, Smoking and Substance Screening Tool (ASSIST) | Change from baseline to 1 week post-program (13 weeks from baseline)
  This 8-item measure screens for use, abuse, and dependence on variety of substances ranging from tobacco and alcohol to cannabis, cocaine, and amphetamines (Humeniuk et al., 2008). It has shown to have high reliability in multiple countries including Zimbabwe (Henry-Edwards et al., 2003). Responses are rated on a Likert scale of 1 to 5, ranging from never to daily use. Scores are summed to distinguish low risk, medium risk, and high risk of developing health or other problems from substance use (ASSIST manual, 2003).
Government grants | Change from baseline to 1 week post-program (13 weeks from baseline)
  The extent of government support grants for each family will be determined based on parental report of the major forms of social security transfers (5-items; Government Housing Subsidy, Old Age Pension, Child Support Grant, Foster Care Grant, Pension, and Disability Grant). A dichotomous variable will be created identifying whether the family received any grants. A separate predictor variable will be created specifically for child-related grants (Delaney, 2008).
Parent Physical Illness | Change from baseline to 1 week post-program (13 weeks from baseline)
  Parental sickness will be measured using items from the Health Systems Trust South African Health Review 2006 (Ijumba and Padarath, 2006) and the South African Demographic and Health Survey (Department of Health and Medical Research Council, 2007) (16-items total). Participants will respond positively or negatively on the presence of chronic illnesses (asthma, epilepsy and diabetes), minor ailments (cold/flu and worms), and acute conditions (pneumonia, diarrhea and burns).
AIDS-related child orphanhood and parental HIV-status and/or AIDS-sickness | Change from baseline to 1 week post-program (13 weeks from baseline)
  This study will use parental reports of the Verbal Autopsy Questionnaire (VA; 18 items) to assess child AIDS-related orphanhood and caregiver AIDS-sickness, as well as other orphanhood causes and other sicknesses (Lopman et al., 2006). The VA has been validated in South Africa with a 76% positive prediction rate, 89% sensitivity, and 93% specificity (Hosegood et al., 2004, Kahn et al., 2000). This study will use a conservative approach requiring the presence of 3 or more AIDS-related symptoms defined by the World Health Organization (e.g. - oral candidiasis, respiratory tract infection, and persistent diarrhea) in order to determine caregiver HIV-status and/or AIDS-related parental mortality (WHO, 1994). To avoid potential stigmatization, items from the VA will be interspersed among items measuring other physical illnesses.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Ward, PhD, Principal Investigator — University of Cape Town; Lucie Cluver, DPhil, Principal Investigator — University of Oxford
Locations (1):
- Ikamva Labantu Wellness Centre, Cape Town, Western Cape, South Africa